CLINICAL TRIAL: NCT04197999
Title: A Phase 1b, Single and Multiple Dose, Open-Label Trial of Intravenous GMI-1359 in HR+ Metastatic Breast Cancer Subjects
Brief Title: A Study to Determine Safety and Tolerability of GMI-1359 in Subjects With HR+ Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After demonstrating the on target effect of GMI-1359 via pharmacodynamic markers (CXCR4 and E-selectin), Sponsor terminated the trial due to COVID-related slow enrollment.
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMI-1359-210
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: HR+ Metastatic Breast Cancer; Breast Cancer; Breast Cancer Metastatic
Keywords: GMI-1359; breast cancer; HR+ metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Ascending Dose followed by Multiple Doses (Experimental): Up to 3 single ascending doses of GMI-1359 followed by the highest tolerated dose given for 3 consecutive days.
  Interventions: Drug: GMI-1359

INTERVENTIONS:
Drug: GMI-1359 — Injection 10 mg/mL

SUMMARY:
This trial is being conducted to investigate the safety, tolerability, pharmacokinetics (the effect the body has on the drug), and pharmacodynamics (the effect the drug has on the body) of GMI-1359 when given with standard-of-care treatment to subjects with HR+ metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HR+ metastatic breast cancer, currently stable or minimally progressive on current endocrine-based therapy.
* Continuing on current endocrine-based therapy with an aromatase inhibitor, selective estrogen receptor degrader, or selective estrogen receptor modulator; and must be medically eligible to remain on this therapy during the treatment period.

Exclusion Criteria:

* Uncontrolled acute life-threatening bacterial, viral, or fungal infection.
* Subjects who are pregnant or breastfeeding
* Concurrent treatment with any cytotoxic chemotherapy agent or other targeted therapies including HER2 targeting therapies
* Currently receiving, or less than 28 days since ending treatment on another investigational drug.
* Clinically significant cardiovascular disease.
* Abnormal liver function.
* Any medical, psychiatric, or other condition which, in the opinion of the investigator, is likely to interfere with trial completion, assessments, or interpretation of trial results, or otherwise would make the subject an inappropriate subject for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Occurrences of dose-limiting toxicities (DLT) including protocol-defined adverse events (AEs)/serious adverse events (SAEs), and/or laboratory abnormalities will be assessed in order to determine recommended phase II dose (Safety and Tolerability) | Up to 4 months

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve [AUC0-t and AUC0-∞] of GMI-1359 | Up to 16 weeks
Maximum plasma concentration [Cmax] of GMI-1359 | Up to 16 weeks
Time to reach maximum plasma concentration [tmax] of GMI-1359 | Up to 16 weeks
Individual estimate of the terminal elimination rate constant [Λz] of GMI-1359 | Up to 16 weeks
Half-life [t1/2] of GMI-1359 | Up to 16 weeks
Total plasma clearance [CL] of GMI-1359 | Up to 16 weeks
Apparent volume of distribution estimated at the terminal phase [Vz] of GMI-1359 | Up to 16 weeks
Pre- and post-dose circulating tumor cells (CTC) enumeration to determine tumor cell mobilization [digital pathology assay] | Up to 16 weeks
Pre-and post-dose CD34+ cell quantification to determine mobilization into peripheral blood [standard flow cytometry] | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Force, DO, Principal Investigator — Duke University; Dorothy A Sipkins, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No